CLINICAL TRIAL: NCT04995315
Title: Pyruvate Kinase Deficiency Global Longitudinal Registry Substudy of Protocol AG348-C-008: Cognition in Participants With Pyruvate Kinase Deficiency
Brief Title: Pyruvate Kinase Deficiency Global Longitudinal Registry Substudy of Protocol AG348-C-008
Status: Completed | Type: Observational
Sponsor: Agios Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: AG348-C-016
Record Dates: First submitted 2021-07-13; First posted 2021-08-06 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Pyruvate Kinase Deficiency
Keywords: Glycolytic enzymopathy; Congenital Nonspherocytic hemolytic anemia (CNSA); PKD
MeSH Terms: conditions — Pyruvate Kinase Deficiency of Red Cells; Anemia, Hemolytic, Congenital Nonspherocytic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- PK Deficiency Diagnosed Participants: Participants will receive online user access to the CBB. Participants will complete 2 CBB assessments on Study Day 0 and Study Day 90.

SUMMARY:
This is a substudy of Study AG348-C-008, an observational, longitudinal, multicenter, global registry that aims to better understand the longitudinal clinical implications of pyruvate kinase deficiency (PK deficiency). The primary purpose of this study is to describe the cognition of participants with PK deficiency, as objectively measured by the Cogstate Brief Battery (CBB).

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥18 years of age;
* Participant must be enrolled in Study AG348-C-008.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with PK deficiency will be enrolled in at least 3 sites also participating in Study AG348-C-008. If any participants are unable to complete the Day 0 CBB assessments, additional participants may be enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2021-07-02 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
Change Over Time in Cogstate Brief Battery (CBB) Scores | Day 0, Day 90
  CBB is a series of brief computerized assessments used to evaluate 4 major cognitive domains: psychomotor speed, attention/vigilance, visual learning, and working memory. If the CBB score falls between -10 to +10, it is considered normal. In Cogstate scoring 0 could be considered as performing in the average range, a negative score means below-average performance, and a positive score means above-average performance. A positive change in scores indicates slightly better performance.

SECONDARY OUTCOMES:
CBB Scores of Participants as Compared to the Scores of Age-Matched Controls | Day 0, Day 90
  CBB is a series of brief computerized assessments used to evaluate 4 major cognitive domains: psychomotor speed, attention/vigilance, visual learning, and working memory. An age-standardized score of ≤-1 on a test will be defined as abnormal. Cognitive impairment on the day of testing will be defined as ≥2 tests with abnormal performance.
Percentage of Participants With Blood Transfusions Affecting Cognition, as Assessed by the Investigator | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Medical Affairs, Study Chair — Agios Pharmaceuticals, Inc.
Locations (3):
- Massachusetts General Hospital, Boston, Massachusetts, United States
- Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan, Italy
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No